CLINICAL TRIAL: NCT07323901
Title: GRAPE-GDM Prospective Comperative Trial - Grape Juice as a Replacement Drink for Gestational Diabetes Screening
Acronym: GRAPE-GDM
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: BNZ-0122-24
Record Dates: First submitted 2025-05-07; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-03

CONDITIONS: Pregnancy - Prenatal Testing
MeSH Terms: interventions — Sugars

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- grape juice (Experimental): Participants: Each participant will undergo both the standard GCT and an alternative GCT using 500 ml of grape juice (containing 50g of sugar).
  Control Group: Each participant serves as her own control by completing both tests in a randomized order.
  Interventions: Other: Participants will consume 500 ml of commercially available grape juice which contains 50g of sugar, serving as an alternative glucose load.

INTERVENTIONS:
Other: Participants will consume 500 ml of commercially available grape juice which contains 50g of sugar, serving as an alternative glucose load. — This study investigates a non-carbonated, natural beverage (grape juice) as an alternative glucose-loading method for gestational diabetes screening. Unlike other studies that have explored alternative carbohydrate sources such as jelly beans or gummy candies-which require chewing and may impact dental health-our study focuses on a readily available liquid alternative that closely mimics the glucose absorption kinetics of the standard 50g glucola drink.

SUMMARY:
Study Type: Observational, prospective, multicenter comparative study

Primary Purpose: The goal of this study is to evaluate whether grape juice can serve as an effective alternative to the standard 50g glucola drink for gestational diabetes screening in pregnant individuals at 24-28 weeks of gestation.

Main Questions:

Can an alternative glucose-loading drink (grape juice) provide comparable blood glucose measurements to the standard GCT? Does grape juice improve patient satisfaction and compliance with gestational diabetes screening?

Comparison Group:

Researchers will compare the standard GCT (50g glucola drink) with the alternative GCT (500 ml grape juice containing 50g sugar). Each participant will undergo both tests, serving as her own control, to assess differences in glucose measurements and patient preferences.

Participant Tasks:

Participants will:

- Undergo two glucose challenge tests (GCT): Standard GCT (50g glucola) at their health maintenance organization (HMO) or hospital.

Alternative GCT (500 ml grape juice) during a scheduled visit or hospitalization.

* Have blood drawn one hour after each test for glucose measurement.
* Complete a questionnaire assessing satisfaction and preference between the two methods.
* Provide follow-up information if they require additional testing (e.g., 100g OGTT).

DETAILED DESCRIPTION:
Study Type: Prospective, observational, multicenter comparative study Primary Purpose: To evaluate whether grape juice can serve as an effective alternative to the standard 50g glucola drink for gestational diabetes screening, with the goal of improving patient compliance and satisfaction.

Participant Population: Pregnant individuals at 24-28 weeks of gestation, undergoing routine glucose challenge testing (GCT). Participants will be recruited from Maternal-Fetal Medicine (MFM) clinics, prenatal maternal wards, and social media outreach.

Main Research Questions:

Can an alternative glucose-loading drink (grape juice) provide comparable blood glucose measurements to the standard GCT? Does grape juice improve patient satisfaction and compliance with gestational diabetes screening?

Study Design & Methods:

Participants: Each participant will undergo both the standard GCT and an alternative GCT using 500 ml of grape juice (containing 50g of sugar).

Control Group: Each participant serves as her own control by completing both tests in a randomized order.

Blood Glucose Measurement: A blood sample will be drawn one hour after ingestion of each drink to compare glucose levels.

Follow-up: If necessary, follow-up phone calls will be conducted to collect results from the standard GCT performed at external clinics.

Outcome Measures:

Primary Outcomes:

Mean difference in blood glucose levels between the standard and alternative GCT.

Proportion of patients with a positive screening result (≥140 mg/dL) for both methods.

Sensitivity, specificity, and predictive values of the alternative GCT compared to the standard test.

Agreement between the two methods using Bland-Altman analysis.

Secondary Outcomes:

Patient satisfaction with both screening methods (measured via a Likert scale). Participant preference between grape juice and glucola. Incidence of adverse events (e.g., nausea, dizziness).

Statistical Analysis:

Pearson's correlation and paired t-tests will assess the agreement between glucose measurements.

ROC analysis will determine the diagnostic performance of the alternative test. Bland-Altman plots will evaluate bias and agreement between the two methods.

Sample Size Calculation:

A minimum of 120 participants is required to detect a clinically significant difference, accounting for attrition.

Recruitment Strategy:

Multicenter Approach: Enrollment from two major hospitals (Bnai Zion and Poria).

Social Media Outreach: Targeted campaigns will inform and recruit participants. Incentives: Participants will receive a complimentary MFM consultation and fetal ultrasound.

Significance:

If grape juice proves to be a viable alternative to the standard GCT, it could improve patient compliance, enhance screening participation, and minimize the discomfort associated with traditional glucose testing.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

Pregnant individuals scheduled for routine GCT at 24-28 weeks. Well-dated pregnancy (confirmed first-trimester ultrasound). Willingness to comply with study protocol.

Exclusion Criteria:

High-risk individuals requiring direct 100g OGTT (e.g., prior GDM, BMI >40, PCOS).

Intolerance to the alternative drink. Gastrointestinal conditions affecting glucose absorption such as active bowel disiease.

Recent corticosteroid administration for fetal lung maturity after standard GCT.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Blood glucose concentration after test beverage | one hour from injestion of the drink
  Venous plasma glucose ( measured at 60 minutes after each beverage

SECONDARY OUTCOMES:
Participant satisfaction with glucose drink | One hour after ingestion of the glucose drink.
  Participant reported satisfaction with the consumed glucose drink, assessed using a 5 point Likert scale ranging from 1 (very dissatisfied) to 5 (very satisfied).
Participant preference for glucose challenge test drink | One hour after ingestion of the glucose drink.
  Participant stated preference for the alternative glucose drink compared with the standard glucose challenge test drink, recorded as a categorical variable (alternative drink preferred, standard drink preferred, no preference).
Adverse events following glucose drink ingestion | One hour after ingestion of the glucose drink.
  Occurrence of self reported adverse events following ingestion of the glucose drink, including nausea and dizziness, recorded as present or absent.

OTHER OUTCOMES:
Gestational age at birth | At delivery
  Gestational age at delivery, measured in completed weeks of gestation, based on best obstetric estimate.
Neonatal birth weight | At birth
  Birth weight of the neonate measured in grams immediately after delivery.
Mode of delivery | At delivery
  Mode of delivery categorized as vaginal delivery or cesarean delivery.

CONTACTS AND LOCATIONS:
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No
De identified individual participant data collected in this study will not be shared outside the study team.